CLINICAL TRIAL: NCT05665842
Title: Effects of Sleep Hygiene Education and Music Practice on Insomnia and Quality of Life in Adolescents
Brief Title: The Effects of Education and Music Practice on Insomnia and Quality of Life
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Pınar Tekcan, Principal Investigator, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ErciyesU.PTekcan1
Record Dates: First submitted 2022-12-09; First posted 2022-12-27 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Music Application Group (Experimental): After explaining the purpose of the study and the way it was applied to the adolescents in the music practice group, the Introductory Characteristics Form for Adolescents, PedsQL and AIQ will be applied.
  After, the predetermined instrumental music will be shared with the adolescents every evening for 15 days via social media by the researcher and participants will be asked to listen to these music. Participants will listen to the instrumental music sent by the researcher for at least 20 minutes every evening during the music application. This whole process will be reminded to the adolescents with messages every evening and they will be asked to listen the music before the normal bedtime (before 23:00 at night). At the end of the music application (after 15 days), the Introductory Characteristics Form for Adolescents, PedsQL and AIQ will be reapplied.
  Interventions: Other: Music Application
- Sleep Hygiene Training Group (Experimental): After explaining the purpose of the study and the way it was applied to the adolescents in the music practice group, the Introductory Characteristics Form for Adolescents, the Pediatric Quality of Life Inventory (PedsQL) and Adolescent Insomnia Questionary (AIQ) will be applied.
  Adolescents in this group will be trained on Zoom for 4 weeks, 2 times a week, for 8 sessions (1 session 40 min). Sleep hygiene training prepared based on expert opinions and literature (Halal & Nunes, 2014; Dinis & Bragança, 2018; İşsever et al., 2021) will be given by the researcher. A Sleep Hygiene Training Booklet will be prepared for use in education and to give to adolescents after education.The Sleep Hygiene training booklet to be prepared will be prepared by the researcher and submitted for expert opinions. Adolescents who received sleep hygiene training will be reapply 15 days after the training, with the PedsQL and AIQ.
  Interventions: Other: Sleep Hygiene Training
- Control Group (No Intervention): No attempt will be made to the adolescents who will be in the control group, and the Introductory Characteristics Form for Adolescents, the Pediatric Quality of Life Inventory (PedsQL) and Adolescent Insomnia Questionary (AIQ) will be applied on the same dates in parallel with the education and music application groups.

INTERVENTIONS:
Other: Music Application — The Introductory Characteristics Form for Adolescents, the PedsQL and AIQ will be applied. After, the predetermined instrumental music will be shared with the adolescents every evening for 15 days via social media by the researcher and participants will be asked to listen to these music. Participants will listen to the instrumental music sent by the researcher for at least 20 minutes every evening during the music application. This whole process will be reminded to the adolescents with messages every evening and they will be asked to listen the music before the normal bedtime (before 23:00 at night). At the end of the music application (after 15 days), the Introductory Characteristics Form for Adolescents, the PedsQL and AIQ will be reapplied. In the music application, the selecting instrumental music will be used. To determine the music, the researcher will be advice received from the TÜMATA and the a music education expert.
  Arms: Music Application Group
Other: Sleep Hygiene Training — After explaining the purpose of the study and the way it was applied to the adolescents in the music practice group, the Introductory Characteristics Form for Adolescents, the Pediatric Quality of Life Inventory (PedsQL) and Adolescent Insomnia Questionary (AIQ) will be applied.
  Adolescents in this group will be trained on Zoom for 4 weeks, 2 times a week, for 8 sessions (1 session 40 min). Sleep hygiene training prepared based on expert opinions and literature (Halal & Nunes, 2014; Dinis & Bragança, 2018; İşsever et al., 2021) will be given by the researcher. A Sleep Hygiene Training Booklet will be prepared for use in education and to give to adolescents after education.The Sleep Hygiene training booklet to be prepared will be prepared by the researcher and submitted for expert opinions. Adolescents who received sleep hygiene training will be reapply 15 days after the training, with the PedsQL and AIQ.
  Arms: Sleep Hygiene Training Group

SUMMARY:
Background: Insomnia is the most common problem among sleep disorders. Approximately 4-39% of the general adolescent population appears to experience clinically classified insomnia. Insomnia in adolescence, when intellectual, physiological, psychological and social changes are intense, deprives adolescents of the attention and cognition needed to play an active role in these exciting and challenging processes. The aim of this study was to evaluate the effect of music practice and sleep hygiene education in adolescents aged 14-18 years with insomnia.

Method: The study will conduct in a randomized controlled experimental design with three groups. The population of the study consists of adolescents aged 14-18, who are studying in Amasya City Center. The sample of the study will be 60 adolescents in the sleep hygiene education group (20), the music practice group (20) and the control group (20). The research will be carried out between September and November 2022.In this study, data will with collect Descriptive Characteristics Form for Adolescents and Their Families, Adolescent Insomnia Questionnaire and Quality of Life Scale for Children.

DETAILED DESCRIPTION:
The type of Research It will be conducted as a randomized controlled experimental study in a pre-test-post-test design to determine the effect of sleep hygiene education and music practice on insomnia and quality of life in 14-18 age group adolescents.

Location and Characteristics of the study Research The second phase of this study, which examines the effects of sleep hygiene education and music practice on sleeplessness and quality of life in adolescents, will be conducted with adolescents aged 14-18 who are studying in high schools in the city center of Amasya Provincial Directorate of National Education in the 2022-2023 academic year.

Population and Sample of the Research The universe of the research is high school 9-12 in the city center affiliated to the Amasya Provincial Directorate of National Education in the 2022-2023 academic year. It will consist of adolescents aged 14-18 who attend their classes. The sample number of this study will be determined with the sample calculation of the known universe. In high schools selected using the random numbers table, students with ALS scores of 15 and above (with high insomnia scores) will be determined by applying ALS to as many students as the calculated sample number. Adolescents who will be included in the experimental research part of the second phase of this study will be selected by a simple random method from students who have high insomnia scores and meet the research criteria. For this purpose, the computer program (randomizer.org) will be used.

In the literature review, no similar studies were found for the subject and age group of this study. However, according to the findings of studies on sleep quality in adolescents (Çağlar, 2020) and the power analysis performed in GPower (effect size = 0.97, impact power = 0.90) the sample size varies between 57 adolescents. In this study, it was decided to have 20 samples in each group according to α=95% confidence level and 90% power. After reaching 20 adolescents in each group, power analysis will be calculated using insomnia scores and it will be decided whether the sample size is sufficient or not.

Although the number of students in high schools on the dates of the second phase of the study is not known at the moment, 8464 students in the 14-18 age group continue their education in 21 high schools in the 2021-2022 academic year.

Application In this study, which examines the effects of sleep hygiene education and music practice on insomnia and quality of life of 14-18-year-old adolescents, intervention and control groups will be studied in a pre-test and post-test design. No intervention will be applied to the control group. To the initiative groups; it was planned to apply music to the students in the 1st group, and sleep hygiene training to the students in the 2nd group.

ELIGIBILITY:
Inclusion Criteria:

* Those between the ages of 14-18,
* Receiving 15 points or more in AOS,
* Having no vision, hearing, or speech problems,
* Able to speak and write Turkish,
* No mental or neurological disability,
* Participating in the training program with the zoom program,
* Smartphone, using social media communication (WhatsApp),
* It was planned to include the adolescents who had the permission of themselves and their parents to participate in the study in the second phase of the study.

Exclusion Criteria:

* Adolescents who want to withdraw from the study at any stage of the study will be excluded from the study.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-19 (Estimated); Primary Completion 2023-03-19 (Estimated); Study Completion 2023-12-19 (Estimated)

PRIMARY OUTCOMES:
Adolescent Insomnia Questionnaire | a day before the music application and sleep hygiene education
  Scores from the scale range from 0 to 52, and the higher the score, the higher the insomnia. The cut-off point of the scale was accepted as 15 points and above.
Adolescent Insomnia Questionnaire | through application and education completion, an average of 1 months
  Scores from the scale range from 0 to 52, and the higher the score, the higher the insomnia. The cut-off point of the scale was accepted as 15 points and above.
Quality of Life Scale for Adolescent Form | a day before the music application and sleep hygiene education
  . Scale items are scored between 25 and 100. The total score obtained from the scale is obtained by taking the arithmetic average of the scores obtained from the scale. The higher the total score obtained from the scale, the higher the health-related quality of life
Quality of Life Scale for Adolescent Form | through application and education completion, an average of 1 months
  . Scale items are scored between 25 and 100. The total score obtained from the scale is obtained by taking the arithmetic average of the scores obtained from the scale. The higher the total score obtained from the scale, the higher the health-related quality of life

IPD SHARING:
Plan to Share IPD: Undecided